CLINICAL TRIAL: NCT04807361
Title: Assessment of Accommodation Behavior in Children Under Myopia Control Treatment (Pilot Study)
Status: Completed | Type: Observational
Sponsor: State University of New York College of Optometry (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Xiaoying Zhu, OD, PhD, MD, MS, FAAO, Assistant Clinical Professor, State University of New York College of Optometry
Other Study IDs: IRBNET ID 1525840
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Accomodation; Biofeedback Training; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- (1) Multifocal soft contact lenses (MFCLs): Assess accommodative function of myopic children wearing MFCLs for myopia control treatment. Accommodative stimulus-response functions and accommodative lags will be determined during one, one hour measurement session for four stimulus distances using an IR video refractometer (PowerRefractor). MFCL subjects will also be tested while wearing SVCL distance corrections for comparison.
  Interventions: Behavioral: Auditory biofeedback traing
- (2) orthokeratology: Assess accommodative function of myopic children wearing Orthokeratology for myopia control treatment.
- (3) low-dose atropine: Assess accommodative function of myopic children using low-dose atropine eye drops for myopia control treatment.
- (4) single vision spectacle correction (control): Assess accommodative function of myopic children wearing single vision spectacle lenses.

INTERVENTIONS:
Behavioral: Auditory biofeedback traing — Subjects who wear MFCLs for myopia control will receive one episode of auditory biofeedback training, and their accommodative responses to various demands (0, 2.5, 3, and 4 D) before and after the training were measured using a power refractor.
  Groups: (1) Multifocal soft contact lenses (MFCLs)

SUMMARY:
This study will examine the accommodative behavior in children undergoing myopia control treatments. A subset of children showing reduced accommodation, known to occur in while wearing multifocal soft contact lenses (MFCL) from previous studies, will undergo auditory biofeedback training to improve the accommodative response and possibly improve treatment efficacy. The results of this study will be used to design a larger clinical trial.

Aim 1 - The accommodation response in myopic children being treated with MFCL for six months or longer, will be determined. The accommodative response data will be collected while the patients are wearing the MFCL and will be compared to the baseline control response when the subjects wear single vision soft contact lenses (SVCL). Additional comparisons will include accommodative measures in untreated myopic children wearing spectacle corrections (unttreated controls), children being treated with ortho-keratology contact lenses, and children treated with low-dose atropine (0.01%, considered not to affect accommodation). How these additional myopia treatments affect the accommodation response has yet to be determined.

Aim 2 - Children treated with MFCL who show reduced accommodative responses will undergo a brief period of auditory biofeedback accommodative training to determine whether the response in children can be improved and how long it can be sustained. Improving the accommodative response in these patients may improve the treatment efficacy by increasing the effect of the positive power addition built into the lenses.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected monocular Snellen visual acuity (VA) ≧ 20/25
* Age 8 - 15 years
* Refractive error spherical equivalent between -0.75 D and -10 D
* Astigmatism ≤ 0.75 D
* Age-appropriate amplitude of accommodation
* No suspected or confirmed eye disease (anamnesis)
* No accommodative or binocular function abnormalities
* Agreement to participate in the study (informed consent of parents, assent of child)
* Children who are currently under myopia control treatment should already be so for ≥ 6 months

Exclusion Criteria:

* Persons who are incapable of giving consent
* Refractive error spherical equivalent < -10 D and > -0.75 D
* Astigmatism > 0.75 D
* Abnormal binocular functions
* Medication affecting accommodative response or causing dry eye

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric population
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Accommodation | Within 4 weeks
  Subjects' accommodative response will be measured using a power refractor

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Bloomfield, PhD, Study Director — State University of New York College of Optometry
Locations (1):
- State University of New York, College of Optometry, Long Beach, New York, United States